CLINICAL TRIAL: NCT03617796
Title: Prognostic Value of CD64 Marker for Patients in Intensive Care Unit
Acronym: CD64
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/CD64-GIBOT/MS
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Systemic Inflammatory Response Syndrome; Intensive Care
Keywords: markers CD64
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood samples for CD64 biomarker measurement will be obtained daily during the patient's hospitalization : 30 microlitre (tube bottom - residual volume)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among patients admitted to the intensive care unit (ICU), early recognition of those with the highest risk of death is of paramount importance. Since clinical judgment is sometimes uncertain biomarkers could provide additional information likely to guide critical illness management. We want to evaluate the prognostic value of leucocyte surface expression of CD64.

Blood samples for CD64 biomarker measurement will be obtained daily during the patient's hospitalization. The primary outcome was all-cause death at D28 after admission

DETAILED DESCRIPTION:
Some local or systemic biological markers, using highly specialized techniques, have an interest that remains quite marginal in routine.

Markers of inflammation generally have elevated concentrations in circulating blood, but these increases are not specific for prognosis. This is the case of pro-inflammatory cytokines (TNF, IL-1, IL-6...)[1, 2] and especially, so-called'acute phase' proteins such as C-reactive protein (CRP) and procalcitonin. It is now well established that the rise in the CRP is totally non-specific. With regard to procalcitonin, the published data are far from univocal[3-4], in particular because of the heterogeneity of the populations studied (emergency services, medical services, intensive care).

These conventional biological assays are therefore not very informative and less efficient than the clinical-biological scores used in routine (SAPSII and SOFA).

An alternative diagnostic approach relies on molecular changes in the cellular compartment of innate immunity. Activation of neutrophil polymorphils (PNN) is the result of the pro/anti-inflammatory cytokinic balance and hormonal cascades In other words, the degree of activation of NNPs can be considered as the barometer of the intensity of any acute inflammatory phenomenon. One of the most specific indicators of a systemic inflammatory response is the increased expression of CD64, a high affinity receptor to the immunoglobulin fragment Fcγ, on the surface of PNNs.

CD64 expression elevation is induced in 4-6 hours by numerous cytokines (G-CSF, IFN- γ[5-7]. Given the very low basal expression level of CD64 (less than 2000 sites per cell) and its rate of elevation in case of inflammation, its determination could prove interesting in demonstrating the inflammatory response and its intensity.

In addition, the measurement of CD64 expression has obvious advantages over other PNN activation markers (such as CD11b, CD18, CD16, CD45RA or CD62L): negligible expression in healthy volunteers; no influence of blood sample manipulation; stable expression for 36 hours on anticoagulated blood.

The other decisive advantage is the standardisation and automation of the measurement (performed in flow cytometry) thanks to a device developed by the LeukoDx company, the ACCELLIX-CD64. This measurement is performed in whole blood (30 to 50µL maximum), and the measurement time is short (26 minutes), which makes it particularly attractive in the context of emergency and resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit

Exclusion Criteria:

* Neutropenia (<500 neutrophils/mm3)
* Treatment by G-CSF or IFN-γ during the week preceding admission to intensive care
* Age < 18 years
* Pregnancy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit for any reason
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2018-12-09 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality at 28 days after admission | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi SIAGHY, Mr, Study Director — CHRU de NANCY
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France